CLINICAL TRIAL: NCT04602468
Title: Real World Clinical Outcomes With Novel Modulator Therapy Combinations in People With CF (RECOVER)
Acronym: RECOVER
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Imperial College London (Other); University College Dublin (Other); University of Limerick (Other); Cystic Fibrosis Registry of Ireland (Other); Erasmus Medical Center (Other); Medizinische Hochschule Brandenburg Theodor Fontane (Other); Queen's University, Belfast (Other); Teagasc (Industry); The Hospital for Sick Children (Other); St. James's Hospital, Ireland (Other); Amsterdam UMC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: RECOVER
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis Liver Disease; Cystic Fibrosis in Children; Adherence, Medication; Cystic Fibrosis Gastrointestinal Disease
MeSH Terms: conditions — Cystic Fibrosis; Medication Adherence | interventions — elexacaftor, ivacaftor, tezacaftor drug combination

STUDY DESIGN:
Intervention Model Description: The decision to implement Kaftrio treatment is made completely independently of the decision to enter the study. The investigators will follow the requirements of the local approved Kaftrio SmPC for the patient management as detailed in the 'special warnings and precautions for use' (e.g. management of hepatic impairment, rash, ophthalmological monitoring, between others), and for the management of interaction with other medicinal products and other forms of interactions. The 12+ cohort will be enrolled first on the basis the drug will be approved for children aged 12 and over first. The 6-11 year cohort will only be enrolled when the license is extended to this age group, and treatment with Kaftrio will only occur in the context of prescription by a physician in compliance with marketing authorization and the SPC.
Who Masked: Participant
Masking Description: No blinding. The decision to implement Kaftrio treatment is made completely independently of the decision to enter the study. Those determined to begin treatment on Kaftrio clinically will undergo eligibility assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard group (Other): The standard testing group will be available for both age cohorts with sites having a predefined recruitment cap for each testing group. The standard testing will involve the following assessments; sweat chloride, LCI, height/weight/BMI, FEV1, airway sampling (micro), FeNO, liver function testing, liver ultrasound, liver examination, stool collection, blood collection, abdominal symptom score, CFQ-R, pharmacy records medication pick up rate, adherence questionnaires, MEMs caps and antibiotic use.
  Interventions: Drug: Kaftrio
- Advanced group (Other): In addition to all elements of the standard testing group, the advanced testing group will undergo: Ultra-low dose spirometry-controlled CT scanning, sputum collection and nasal lavage collection. This will be available for both age cohorts with sites having a predefined recruitment cap for each testing group.
  Interventions: Drug: Kaftrio

INTERVENTIONS:
Drug: Kaftrio — The intervention is the same for both study groups. In addition to all the assessments in the standard arm, the advanced arm subjects will undergo spirometry controlled CT, nasal lavage and sputum sample collection.
  Other Names: Trikafta

SUMMARY:
RECOVER is a prospective, multicenter observational study designed to measure the real world clinical effectiveness of elexacaftor, tezacaftor and ivacaftor triple combination therapy (Kaftrio) in people with cystic fibrosis over a two year period. Measured outcomes include measures of lung function, lung inflammation, lung imaging, abdominal symptoms, gut inflammation, liver function, pancreatic exocrine function, nasal inflammation, quality of life and adherence to therapy. The study will examine outcomes in children aged six years and above over a period of two years. The first phase of the study will commence in 2020, recruiting children 12 years and older who have started on clinical treatment with Kaftrio.

DETAILED DESCRIPTION:
Our aim with RECOVER is to examine the clinical impact of Kaftrio on key clinical outcomes in people with CF in a real-world setting. For this study, in addition to some of the more traditional ways of monitoring clinical outcomes in people with CF such a standard lung function, nutrition, exacerbations and liver disease, we are proposing to include some novel outcome measures not typically used in clinical trials such as lung clearance index (LCI) and spirometry controlled chest CT.

By implementing an extensive study protocol that will include important outcomes in a number of areas of health in people with CF, and matching this to a comprehensive biosample collection plan, we will have the power to gain important insight into how Kaftrio works, and what impact it has on rescue of CFTR function in this group of people.

Data on the following outcomes will be collected during the study:

Lung Clearance Index Ultra-low dose, spirometry-controlled CT scanning Sweat Chloride Nasal Lavage (inflammatory markers and microbiome) Fraction of Exhaled Nitric Oxide (FeNO) Liver Ultrasound Liver examination (signs of liver disease) Sputum Collection (inflammatory markers and microbiome) Stool Collection (inflammation, microbiome, fecal elastase) Abdominal symptom questionnaire CFQ-R (quality of life) Adherence to treatment Height, weight, BMI Forced Expiratory volume in 1 second (FEV1) Microbiological culture of airway specimens (clinical laboratories at sites)

The Lead Investigator is Paul McNally, with Prof. Jane Davies as Co-Lead Investigator. The study will operate in collaboration with our academic and clinical partners and the CF registries in Ireland and the UK. The study is supported by the European CF Society Clinical Trials Network (ECFS-CTN). The study is being run as a CTIMP in the UK clinical sites, as determined by the MHRA. In the Irish sites, the HPRA has determined this study to be an observational research study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria People with CF aged 12 years and over: Participants may only be selected for inclusion in RECOVER if they have been independently determined by their treating physician to be suitable for treatment with Kaftrio in compliance with the official marketing authorization and summary of product characteristics (SPC). The decision to include participants in the study is independent of decision to prescribe Kaftrio. Participants will receive treatment only through prescription by their physician through usual clinical treatment pathways.

Children aged 6-11 years: Children aged 6-11 years will be included in the study only if and when Kaftrio is licenced, approved and funded for this age group. Participants may only be selected for inclusion in RECOVER if they have been independently determined by their treating physician to be suitable for treatment with Kaftrio in compliance with the official marketing authorization and summary of product characteristics (SPC). The decision to include participants in the study is independent of decision to prescribe Kaftrio. Participants will receive treatment only through prescription by their physician through usual clinical treatment pathways.

Subjects on Kaftrio In exceptional circumstances where baseline clinical data has been collected prior to the start of treatment either through clinical care or ethically approved research projects (including a cohort of subjects initially recruited to this study on the understanding that it was a non-regulated observational study) subjects already receiving Kaftrio may be recruited to this study and undergo on-treatment visits. Any additional patient data can only be added with written informed consent from the patients/parents concerned.

All Subjects (people with CF aged 12 years and over, children aged 6-11 years and subjects on Kaftrio) must be taking the full dose of Kaftrio (in accordance with the age appropriate posology in the SmPC).

All subjects must have a signed informed consent form and/or signed assent form when appropriate, as determined by the subjects age and individual site and country standards.

Male and female participants of childbearing potential must agree to adhere to contraception requirements as detailed in the local Kaftrio SmPC and in line with the standard of care.

Exclusion Criteria:

Patients not willing to comply with study procedures or assessments.

Individuals on clinical trials of investigational CFTR modulators.

Clinical instability at baseline assessments. Subjects undergoing an active exacerbation and at the beginning of their treatment should be excluded from the study as this is likely to skew the data.

Any contraindication to Katrio treatment as per the local approved SmPC.

Severe hepatic impairment.

Pregnant and breastfeeding women.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of treatment with TCMT on pulmonary function (FEV1 and LCI) in children and adults with CF over a period of 2 years. | 24 month period
  Spirometry, LCI

SECONDARY OUTCOMES:
To determine the effect of treatment with TCMT on spirometry-controlled CT scores in children and adults with CF over a two-year period. | 24 month period
  Spirometry controlled CT
To determine the effect of treatment with TCMT on airway infection and inflammation in children and adults with CF | 24 month period
  Sputum sample collection, Nasal lavage, airway sampling (microbiology), Sinus sypmptoms (CFQ-R), FeNO
To determine the effect of treatment with TCMT on nutrition, gastrointestinal symptoms, gut inflammation and pancreatic function in children and adults with CF over a two-year period | 24 month period
  Abdominal symptom questionnaire, fecal sample, liver examination, liver ultrasound, liver function tests
To determine the effect of treatment with TCMT on antibiotic treatment of pulmonary disease in children and adults with CF over a two-year period | 24 month period
  Medication possession ratio (MPR)
To assess the impact of the introduction of TCMT on adherence with overall medical treatments for CF | 24 month period
  MEMs caps, adherence questionnaires, Medication possession ratio (MPR)

CONTACTS AND LOCATIONS:
Locations (7):
- Ireland (5):
  - Children's Health Ireland at Crumlin, Dublin, Leinster
  - Children's Health Ireland at Temple Street, Dublin
  - St. Vincent's University Hospital, Dublin
  - University Hospital Limerick, Limerick
  - Children's Health Ireland at Tallaght, Tallaght
- United Kingdom (2):
  - Royal Belfast Hospital for Sick Children, Belfast
  - Royal Brompton Hospital, London

REFERENCES:
- [Derived] McNally P, Lester K, Stone G, Elnazir B, Williamson M, Cox D, Linnane B, Kirwan L, Rea D, O'Regan P, Semple T, Saunders C, Tiddens HAWM, McKone E, Davies JC; RECOVER Study Group. Improvement in Lung Clearance Index and Chest Computed Tomography Scores with Elexacaftor/Tezacaftor/Ivacaftor Treatment in People with Cystic Fibrosis Aged 12 Years and Older - The RECOVER Trial. Am J Respir Crit Care Med. 2023 Nov 1;208(9):917-929. doi: 10.1164/rccm.202308-1317OC. PMID 37703083
- See also: RCOVER Study website — https://recovercf.ie/
- See also: RECOVER Twitter Account — https://twitter.com/StudyCf